CLINICAL TRIAL: NCT05775380
Title: The Role of Pioglitazone in Vascular Transcriptional Remodeling in Individuals Undergoing Coronary Artery Bypass Grafting
Brief Title: The Role of Pioglitazone in Vascular Transcriptional Remodeling
Acronym: PREVALENT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Andrei Carvalho Sposito, Professor of cardiology, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PREVALENT
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Myocardial Reperfusion Injury
MeSH Terms: conditions — Myocardial Reperfusion Injury | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pioglitazone (Active Comparator): Research participants will be randomized to receive pioglitazone hydrochloride 45mg/day for 5 days prior to coronary artery bypass surgery.
  Interventions: Drug: Pioglitazone 45 mg
- Placebo (No Intervention): Research participants will be randomized to not receive intervention in the days prior to coronary artery bypass graft surgery.

INTERVENTIONS:
Drug: Pioglitazone 45 mg — We investigated the role of pioglitazone hydrochloride 45mg/day for five days in patients admitted for coronary artery bypass grafting (CABG) in order to investigate vascular SPhk1 expression, vascular transcriptome and proteome remodeling, as well as S1P content in HDL
  Other Names: pioglitazone hydrochloride
  Arms: Pioglitazone

SUMMARY:
Acute myocardial infarction (AMI) remains the leading cause of death worldwide. In this scenario, early coronary reperfusion is the main therapeutic strategy as it substantially reduces mortality. Paradoxically, however, reperfusion triggers additional tissue damage that accounts for about 50% of the infarcted heart mass, i.e., ischemia and reperfusion injury (IRL). In this context, sphingosine-1-phosphate (S1P) is a sphingolipid synthesized by sphingosine kinases (Sphk), carried in plasma bound to high-density lipoprotein (HDL) and released after cellular damage such as LIR. Particularly, in animal models of AMI, therapies targeting downstream S1P receptor signaling triggered by HDL/S1P are able to promote endothelial barrier functions and attenuate secondary damage to LIR. Thus, the molecular control of sphingosine kinase 1 (Sphk1) transcription during LIR in vivo or during hypoxia/reoxygenation (H/R) in vitro may represent an important mechanism for maintaining endothelial homeostasis since it promotes the generation of S1P and this may promote subsequent HDL enrichment. Thus, the role of pioglitazone hydrochloride 45mg/day for five days in volunteers undergoing coronary artery bypass grafting (BVR) will be investigated in order to verify the vascular expression of SPhk1, transcriptome and vascular proteome remodeling, as well as S1P content in HDL.

DETAILED DESCRIPTION:
This will be a prospective, randomized and open clinical study. From a sample of patients hospitalized for myocardial revascularization surgery, followed at the cardiac surgery outpatient clinic, 20 research participants, male, aged over 40 years, non-diabetic or diabetic with disease duration of less than 10 years, glycated hemoglobin <8% and non-user of NPH insulin, body mass index (BMI) between 20 and 34.9kg/m2 and glomerular filtration rate above 45mL/min who will be monitored at the Hospital de Clínicas/UNICAMP and randomized to receive pioglitazone hydrochloride 45mg/day for 5 days before surgery. The amount of S1P in HDL at baseline (before surgery) will be assessed. This same measurement will be repeated on day 5 (coinciding with the day of surgery) after using pioglitazone hydrochloride 45mg/day. In addition, on the day of surgery, a saphenous vein fragment of approximately 2 cm and an internal thoracic artery fragment of approximately 1 cm will be collected, which will not impair the quality of the graft nor the extent of the material to be used as a graft, because in this case the vascular material is abundant. An aortic artery button and an atrial appendage button will also be collected, which will be discarded. In addition, the results of serum troponin levels in the first 24h post-SVR (6, 12, 24h) will be evaluated to estimate the extent of troponin release. Postoperative examination.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals
* Individuals undergoing CABG surgery for coronary artery disease
* Be over 40 years of age
* BMI between 20 and 34.9kg/m2
* Non-diabetic or if diabetic, disease duration < 10 years, Hba1c < 8%, non-user of NPH insulin
* Ejection fraction > 40%
* Glomerular filtration rate > 45 mL/min

Exclusion Criteria:

* BMI greater than 35 kg/m2, steatohepatitis, chronic kidney disease, systemic vasculitis, conditions that induce systemic inflammation such as psoriasis and systemic lupus erythematosus
* contraindications to the use of pioglitazone hydrochloride (heart failure, liver failure - AST or ALT > 2.5x upper normal limit, history of bladder cancer or macroscopic hematuria without investigation)
* moderate or severe valve disease
* need for concomitant use of other hypoglycemic therapies during hospitalization, particularly insulin
* peripheral edema
* recent hospitalization
* known allergy to any study drug
* polyuria, polydipsia, weight loss, or other clinical signs of volume depletion or diabetes, difficult-to-control systemic arterial hypertension, defined as individuals taking 4 or more drugs
* those who withdraw the Informed Consent Form (TCLE), or who, for some reason, are not able to sign or understand the TCLE
* history of gastrointestinal disorders that may interfere with study drug absorption
* research participant who is participating in other clinical trials or whose participation ended less than six months ago
* Research participant who has left ventricular dysfunction

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-12-22 (Estimated)

PRIMARY OUTCOMES:
HDL-S1P change | Five days
  Change in S1P content of isolated HDL between baseline and after treatment with pioglitazone hydrochloride 45 mg/day

SECONDARY OUTCOMES:
SPHK1 - internal thoracic artery | Five days
  Difference in SPHK1 expression in the internal thoracic artery cells determined by western blot between groups
S1PR1 - saphenous vein | Five days
  Difference in S1P receptor (S1PR1) expression in saphenous vein endothelial cells determined by western blot between groups
SPHK1 - aortic artery | Five days
  Difference in SPHK1 expression in the aortic artery cells determined by western blot between groups;
SPHK1 - atrial appendage | Five days
  Difference in SPHK1 expression in the atrial appendage cells determined by western blot between groups;

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Sposito, Professor, Principal Investigator — University of Campinas, Brazil
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No